CLINICAL TRIAL: NCT06703788
Title: Establishing a Traditional Chinese Medicine Day Care Program for the Prevention and Treatment of Metabolic Syndrome
Brief Title: Integrated Traditional Chinese Medicine Day Care Program for Metabolic Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Principal Investigator, Hsing-Yu Chen, MD, Professor, Chang Gung Medical Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOHW113-CMAP-M-113-000003-B
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Metabolic Syndrome; Dyslipidemias; Diabetes Mellitus
Keywords: obesity; metabolic syndrome; dyslipidemia; diabetes mellitus; integrated traditional Chinese medicine care program
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Dyslipidemias; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Subjects with compatible with diagnosis of metabolic syndrome are the target of this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Integrated traditional Chinese medicine care program (Experimental): Integrated traditional Chinese medicine (TCM) care program for metabolic syndrome, including herbal medicine, laser acupuncture, and diet and lifestyle education based on TCM theory.
  Interventions: Drug: A fiixed combination of Chinese herbal medicine; Device: Laser acupuncture

INTERVENTIONS:
Drug: A fiixed combination of Chinese herbal medicine — a fixed combination of Chinese herbal medicine with Ma-Xing-Gang-Shi-Tang (initiate at 2 grams, with increments of 0.5 grams every 2-4 weeks, up to a maximum dose of 4 grams once daily) and Coptis chinensis (initiate at 0.5 grams, with increments of 0.5 grams every 2-4 weeks, up to a maximum dose of 1 gram once daily), twice a day
Device: Laser acupuncture — Laser acupuncture could be used based on medication therapy at following acupoints: CV9, ST25, SP15, ST28, ST40, and two auricular points (stomach and hunger points)

SUMMARY:
The goal of this study is to evaluate if a integrated tradtional Chinese medicine (TCM) program for improving metabolic syndrome is applicable. It will also learn about the importance of gut microbiome of subjects with ineffective management. The main questions it aims to answer are:

Does a integrated tradtional Chinese medicine (TCM) program could improve metabolic syndrome in six months? Researchers will also explore the determinant factors of successful improvement in metabolic syndrome, including gut microbiome, life style, TCM management compliance.

Participants will:

Receive integrated TCM program for managing metabolic syndrome. Visit the clinic once every 2-4 weeks for checkups and tests Keep a diary of diet and life style

DETAILED DESCRIPTION:
Metabolic syndrome, as one of the major diseases of modern civilization, significantly impacts cardiovascular, cerebrovascular diseases, and cancer, necessitating interdisciplinary collaboration for its prevention and treatment. Currently, the "National Health Insurance Metabolic Syndrome Prevention and Treatment Program" provides health education and consultation services, but these are limited to the field of Western medicine. Our research team's previous studies have found a correlation between Chinese medicine constitution and leptin levels, demonstrating the unique value of Chinese medicine in personalized health education and dietary recommendations. In terms of medication, a variety of drugs are available to control hyperlipidemia, hypertension, and hyperglycemia, but for patients in the early stages of metabolic syndrome, exercise and dietary adjustments remain the primary methods. Obesity and its related complications impose significant economic burdens on both society and individuals. Currently, the main methods of treating obesity include lifestyle adjustments, pharmacological interventions, and weight-loss surgery. However, these methods present challenges in maintenance, medication risks, and side effects. This study also considers the potential value of Chinese herbal medicine and laser acupuncture, aiming to assess their role in the prevention and treatment of metabolic syndrome. Retrospective studies have shown that various Chinese herbs are effective in weight reduction and improving metabolic indicators, and laser acupuncture has shown promise as a method of weight reduction.

The project's objectives include expert meetings to explore models of Chinese medicine in the management of metabolic syndrome to discuss the healthcare models of TCM in the prevention and treatment of metabolic syndrome in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 to 75 years who are eligible for health insurance. (Required)

Additional Criteria (Any one of the following):

2-1. Central Obesity: Waist circumference ≥90 cm for men or ≥80 cm for women. 2-2. Elevated blood glucose levels (≥100mg/dL or currently on medication control) 2-3. Elevated blood pressure (systolic pressure ≥130mmHg, diastolic pressure ≥85mmHg, or currently on medication control) 2-4. Elevated triglycerides (≥150mg/dL, or currently on medication control).High-Density Lipoprotein Cholesterol (HDL-C) < 40mg/dL for men or < 50mg/dL for women, or currently on medication) 2-5. Obesity: BMI ≥ 37.5 or BMI ≥ 32.5 with high-risk complications, such as type 2 diabetes mellitus with glycated hemoglobin levels remaining above 7.5% despite medical treatment, hypertension, sleep apnea syndrome, or fatty liver.

Exclusion Criteria:

* 1. Pregnant or breast-feeding women 2. Endocrine disorders (uncontrolled hypo/hyperthyroidism, adrenal gland disorder) 3. Diagnosis of neurologic or psychiatric diseases 4. Liver or renal dysfunction (AST/ALT higher than 3 times of upper normal limits; eGFR < 60 mL/min/1.73 m2) 5. Acute stress condition (severe infection, receive major surgery in the recent 1 month) 6. Vision, or hearing impairment 7. With other clinical trial medication 8. With Chinese herbal medicine, acupuncture, electroacupuncture or other traditional Chinese medicine (TCM) managements for obesity or metabolic syndrome in the recent 1 month 9. Heavy smoker, alcoholism or substance abuse 10. Severe organ dysfunction: malignancies, autoimmune diseases

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The composite metabolic endpoint | From date of enrollment until the date of end of study. Follow up parameters every one month, up to six months.
  Body mass index (BMI) decrease one point (or body weight decrease at least 5% from baseline), waist circumstance decrease at least 3%, the glycated haemoglobin decrease at least 10% or lower than 5.7%, blood pressure <130/80 mmHg, low-density lipoprotein cholesterol <130 mg/dl and triglyceride <150mg/dL will be used as composite metabolic outcome. Meet any of the above criteria is considered achieving the treatment goal.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan and Linkou branches, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data sharing would be done upon adequate request and approval from the IRB committee of the Chang Gung Medical Foundation.

REFERENCES:
- [Background] Liao YN, Chen HY, Yang CW, Lee PW, Hsu CY, Huang YT, Yang TH. Chinese herbal medicine is associated with higher body weight reduction than liraglutide among the obese population: A real-world comparative cohort study. Front Pharmacol. 2022 Sep 9;13:978814. doi: 10.3389/fphar.2022.978814. eCollection 2022. PMID 36160410
- [Background] Yu WL, Liao YN, Yang TH, Yang CW, Kao TI, Lee PW, Hsu CY, Huang JL, Huang YT, Chen HY. Laser Acupuncture versus Liraglutide in Treatment of Obesity: A Multi-Institutional Retrospective Cohort Study. Healthcare (Basel). 2024 Jun 26;12(13):1279. doi: 10.3390/healthcare12131279. PMID 38998814